CLINICAL TRIAL: NCT02937324
Title: The CloudUPDRS Smartphone Software in Parkinson's Study - a Pilot Dual-site, Open Label Study Comparing the Validity of Smartphone Software for Monitoring the Symptoms and Signs of Parkinson's Disease.
Brief Title: The CloudUPDRS Smartphone Software in Parkinson's Study.
Acronym: CUSSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 16/0062
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2018-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical Assessment (Active Comparator): Motor assessment will be performed by a clinician using the Unified Parkinson's Disease Rating Scale.
  Interventions: Other: Clinical assessment
- Smartphone assessment (Experimental): CloudUPDRS smartphone software assessment will be performed.
  Interventions: Device: CloudUPDRS smartphone software assessment

INTERVENTIONS:
Device: CloudUPDRS smartphone software assessment — Smartphone software consisting of a series of tapping and tremor-measurement tests designed to measure a subset of the UPDRS.
  Arms: Smartphone assessment
Other: Clinical assessment — A clinician will assess the motor signs of the participant using the Unified Parkinson's Disease Rating Scale. The examination will be videoed and rated by 3 blinded examiners.
  Arms: Clinical Assessment

SUMMARY:
This study compares the validity and usability of smartphone software for home monitoring of symptoms and signs in Parkinson's disease as compared to the current clinical gold standard - the Unified Parkinsons Disease Rating Scale.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a neurodegenerative condition, which when treated can result in fluctuating motor activity - sometimes too much movement, sometimes too little.

A series of tests, run on a smartphone, will be used to evaluate the motor signs of Parkinson's and related to a clinical evaluation based on the Unified Parkinson's Disease Rating Scale. 60 participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with probable idiopathic Parkinson's Disease according to Brain Bank criteria (Gibb and Lees, 1988).
2. Over 18 years old.
3. Achieve >20/30 on the Montreal Cognitive Assessment (MOCA).
4. They must have been on the current Parkinson's Disease medication schedule for at least a week and have no plans to change this during the period of testing.
5. They must have the capacity to consent to take part in the study.
6. They must be able to understand English to the level of being able to operate the phone software, follow its instructions and be able to answer the study questions.

Exclusion Criteria:

1. Acute medical illness.
2. Any other co-morbidity that in the opinion of the Investigator may preclude their participation in the study.
3. Unable to consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Validity of smartphone software for home monitoring in Parkinson's disease | 3 years
  The primary objective is to measure the validity (bias and reliability) of the smartphone UPDRS (smartphone derived UPDRS). The primary objective outcome measure is the accuracy (and error) of the smartphone UPDRS predictions of the clinical UPDRS rating score. This will be ascertained by using multiple cross-validation runs in which the data are randomly split into 'calibration' and 'testing' cohorts. The model will be trained on the 'calibration' dataset, and the accuracy and error from the out-of-sample predictions will be summarised into a mean accuracy and error score.

OTHER OUTCOMES:
Data exploration | 3years
  Data from this study will be subjected to post hoc analysis to explore future hypotheses in this area.

CONTACTS AND LOCATIONS:
Overall Officials: Kailash Bhatia, MD, Principal Investigator — University College, London
Locations (1):
- Ashwani Jha, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No